CLINICAL TRIAL: NCT06252506
Title: Molecular Imaging Study of Harmine/DMT: a Basic Research Approach
Acronym: HaD-PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HaD-PET; 320030_204978 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neuropharmacological Investigation of Ayahuasca Constituents DMT and Harmine
Keywords: Brain; Glucose; PET; FDG; Metabolism; DMT; Harmine; Ayahuasca
MeSH Terms: interventions — N,N-Dimethyltryptamine; Harmine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo first, intervention second (Experimental): Participants allocated to this arm receive placebo on their first study day and the active drug under investigation on the second study day.
  Interventions: Drug: N,N-dimethyltryptamine (DMT) + harmine; Drug: Placebo
- Intervention first, placebo second (Experimental): Participants allocated to this arm receive the active drug under investigation on their first study day and placebo on the second study day.
  Interventions: Drug: N,N-dimethyltryptamine (DMT) + harmine; Drug: Placebo

INTERVENTIONS:
Drug: N,N-dimethyltryptamine (DMT) + harmine — DMT and harmine are the two most abundant chemicals in the Amazonian hallucinogenic plant brew, Ayahuasca, which is used traditionally in spiritual and healing ceremonies. An oral formulation of these two substances will be tested against placebo in the context of an FDG-PET scan.
Drug: Placebo — Placebo will be administered on one of the study days to compare the effects of DMT and harmine with the effects a placebo administration.

SUMMARY:
The few reports on effects of psychedelic substances on cerebral metabolic rate (CMRglc) indicate increases (psilocybin; human FDG-PET) or decreases (LSD, rat autoradiography; 5-MeO-DMT rat autoradiography). There are no reports of effects of DMT and/or harmine on cerebral energy metabolism. The primary objective of this study is thus to assess acute cerebrometabolic effects of harmine/DMT in healthy volunteers using quantitative FDG-PET, that is, to measure CMRglc before and after simultaneous treatment with an oral harmine and DMT formulation developed (and already applied) by the investigators' project partners at the University of Zurich. As a secondary objective, the researchers aim to correlate the time-dependent effects on CMRglc as assessed in the PET images with the time-dependent self-reported intensity of participants' psychedelic experience.

ELIGIBILITY:
Inclusion Criteria:

* Between 25-45 years old
* Good command of the German language
* Willing and capable to give consent for the participation in the study after it has been thoroughly explained
* Willing and capable to comply with all study requirements
* Body mass index (BMI) between 18.5 and 35
* Previous experience with psychedelics, but not in the past three months
* Willing to abstain from alcohol, caffeinated drinks, nicotine, food, and sugary drinks for two hours prior to the PET scan on the testing day, and from consuming psychoactive substances for 2 weeks before the first testing day and for the duration of the study

Exclusion Criteria:

* Previous significant adverse response to a psychedelic drug
* Recent or concurrent participation in another study where pharmaceutical compounds will be given
* Presence of Axis I affective, anxiety, or dissociative disorders
* Present or antecedent diagnosis of bipolar disorder (I, II, not otherwise specified), schizophrenia, schizoaffective disorder, psychosis, or other disorders from the psychotic spectrum
* First-degree relatives with present or antecedent schizophrenia, schizoaffective disorder, or bipolar disorder type I
* History of head trauma, seizures, cancer, or cerebrovascular accidents
* Recent cardiac or brain surgery
* Current abuse of medication or psychotropic substances according to SCID I criteria
* Presence of major internal or neurological disorders (including sepsis, pheochromocytoma, thyrotoxicosis, drug-induced fibrosis, familiar or basilar artery migraine)
* Cardiovascular disease (hypertonia, coronary artery disease, heart insufficiency, myocardial infarction, coronary spastic angina) Version 5, 15/11/2023 16/44
* Peripheral vascular disease (thromboangiitis obliterans, luetic arteritis, severe arteriosclerosis, thrombophlebitis, Raynaud's disease)
* Cerebrovascular disease (e.g., stroke, intracranial bleeding / hemorrhage, intracranial aneurysm)
* Diabetes Type 1/2, Metabolic Syndrome
* Serious abnormalities in ECG or blood count/chemistry
* Liver or renal or pulmonary disease
* Inability to lie still in the scanner for about 90 minutes (e.g., because of sneezing, itching, tremor, pain)
* Left-handedness
* Significant radiation exposure (either X-ray or nuclear medicine studies) in the last 12 months
* Presence of claustrophobia or other contraindications to PET scanning
* Presence of contraindications to MRI investigations: Magnetic parts in the body (piercings, brain aneurysm clip, implanted neural stimulator/cardiac pacemaker/defibrillator/Swan Ganz catheter/insulin pump, cochlear implant); metal shrapnel or bullet, ocular foreign body (e.g., metal shavings); current or previous job in metalworking industry
* Current use of medications with significant interaction potential with MAO inhibitors (e.g., antidepressants, antipsychotics, psychostimulants, dopaminergic/serotonergic agents, anticonvulsants)
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, serious current stressors, lack of social support).

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cerebral metabolic rate for glucose (CMRglc) | From enrollment to the second PET scan, up to 6 months
  Differences in CMRglc during a placebo PET scan vs. active-drug PET scan are measured.

SECONDARY OUTCOMES:
Blood Glucose levels | From enrollment to the second PET scan, up to 6 months
  Glucose levels in blood are measured before and after PET scans to correct PET data to changes in glucose during the scans.
Plasma concentrations of DMT, harmine, and their metabolites | From enrollment to the second PET scan, up to 6 months
  Plasma concentrations of DMT, harmine and their main metabolites are assessed at several timepoints, i.e. at baseline, 20, 40, 60, 80, 100, and 180 min after drug or placebo administration. These concentrations serve as a combined outcome measure, as harmine directly influences the metabolism of DMT.
Aliveness Task | From enrollment to the second PET scan to a maximum of 6 months
  Behavioral experiment designed to assess the attribution of consciousness and intentionality to animate and inanimate objects.
Acute Subjective Effects | From enrollment to the second PET scan, up to 6 months
  Acute substance effects are measured with a questionnaire named APsych and consists of 8 items (i.e. ratings of intensity, challenging, acceptance, clarity, visual hallucinations, emotionality, liking, arousal) rated from 1-10 with 10 being the highest and assessment if bodily or psychiatric symptoms are present are assessed at several timepoints, i.e. at baseline, 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, and 300 min after drug or placebo administration.
Blood pressure | From enrollment to the second PET scan, up to 6 months
  Blood pressure is assessed at several timepoints, i.e. at baseline, 20, 40, 80, 180, and 300 min after drug or placebo administration.
Heart rate | From enrollment to the second PET scan, up to 6 months
  Heart rate is assessed at several timepoints, i.e. at baseline, 20, 40, 80, 180, and 300 min after drug or placebo administration.
Challenging Experiences | From enrollment to the second PET scan, up to 6 months
  Challenging Experiences Questionnaire is administered 240 min after drug or placebo administration. The questionnaire consists of 26 items that are rated from 0 (not at all) to 5 (extreme).
Mystical Experience | From enrollment to the second PET scan, up to 6 months
  Mystical Experience Questionnaire is administered 240 min after drug or placebo administration. The questionnaire consists of 30 items that are rated from 0 (not at all) to 5 (extreme).
Emotional Breakthrough | From enrollment to the second PET scan, up to 6 months
  Emotional Breakthrough Inventory is administered 240 min after drug or placebo administration. The questionnaire consists of 6 items that are rated from 0 (not at all) to 100 (very much).
Altered States of Consciousness | From enrollment to the second PET scan, up to 6 months
  Altered States of Consciousness Questionnaire is administered 240 min after drug or placebo administration. The questionnaire consists of 94 items that are rated from 0 (no, not more than usual) to 100 (yes, much more than usual).
Attribution of Consciousness Questionnaire | From enrollment to the second PET scan, up to 6 months
  The Attribution of Consciousness Questionnaire is assessed at baseline (medical screening) and 240 min after drug or placebo administration. The questionnaire consists of 10 items that are rated from 0 (strongly disagree) to 6 (strongly agree).
Individual Differences in Anthropomorphism | From enrollment to the second PET scan, up to 6 months
  The Individual Differences in Anthropomorphism Questionnaire is assessed at baseline (medical screening) and 240 min after drug or placebo administration. The questionnaire consists of 30 items that are rated from 0 (not at all) to 10 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Cumming, PhD, Principal Investigator — Insel Group AG
Locations (2):
- Switzerland (2):
  - Department of Nuclear Medicine, Bern University Hospital, Bern
  - Psychiatric University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vollenweider FX, Leenders KL, Scharfetter C, Maguire P, Stadelmann O, Angst J. Positron emission tomography and fluorodeoxyglucose studies of metabolic hyperfrontality and psychopathology in the psilocybin model of psychosis. Neuropsychopharmacology. 1997 May;16(5):357-72. doi: 10.1016/S0893-133X(96)00246-1. PMID 9109107
- [Background] Berlowitz I, Egger K, Cumming P. Monoamine Oxidase Inhibition by Plant-Derived beta-Carbolines; Implications for the Psychopharmacology of Tobacco and Ayahuasca. Front Pharmacol. 2022 May 2;13:886408. doi: 10.3389/fphar.2022.886408. eCollection 2022. PMID 35600851
- [Background] Egger K, Gudmundsen F, Jessen NS, Baun C, Poetzsch SN, Shalgunov V, Herth MM, Quednow BB, Martin-Soelch C, Dornbierer D, Scheidegger M, Cumming P, Palner M. A pilot study of cerebral metabolism and serotonin 5-HT2A receptor occupancy in rats treated with the psychedelic tryptamine DMT in conjunction with the MAO inhibitor harmine. Front Pharmacol. 2023 Sep 28;14:1140656. doi: 10.3389/fphar.2023.1140656. eCollection 2023. PMID 37841918